CLINICAL TRIAL: NCT06594588
Title: Individualized Exploration of Aerobic Exercise-assisted Treatment of Depression Monitored by Smart Band: a Randomized Controlled Trial
Brief Title: Individualized Exploration of Aerobic Exercise-assisted Treatment of Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Weihua Yue, Professor, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-11
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Depression - Major Depressive Disorder
Keywords: Aerobic exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic exercise group (Experimental): Aerobic exercise intervention combined with conventional drug treatment
  Interventions: Behavioral: Aerobic exercise
- Waiting control group (No Intervention): Antidepressants were routinely used and aerobic exercise interventions were performed at the end of the 8-week follow-up

INTERVENTIONS:
Behavioral: Aerobic exercise — Moderate-intensity aerobic exercise for 30-50 minutes three times a week was added to usual medical therapy
  Arms: Aerobic exercise group

SUMMARY:
The goal of this project is to quantify the relative effectiveness of aerobic exercise monitored by smart wristbands in assisting the treatment of depression and improving cognitive function. It aims to explore the mechanisms through which aerobic exercise exerts its effects using imaging genetics and other methods, and to identify suitable populations for exercise, ultimately providing personalized clinical exercise prescriptions. This study will intervene from a behavioral perspective and also seeks to motivate participants to change and improve their physical activity habits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-45 years (including 18 and 45), no gender restriction;
2. Meets the diagnostic criteria for depressive disorders according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V);
3. Outpatients or inpatients; Hamilton Depression Rating Scale 17-item (HAMD-17) score ≥ 14; Mood Disorder Questionnaire (MDQ) screening negative to exclude bipolar disorder patients; and Clinical Global Impressions-Severity (CGI-S) score ≥ 4;
4. Maintained on antidepressant treatment for at least 4 weeks or not using antidepressant treatment;
5. Written informed consent obtained from the patient.

Exclusion Criteria:

1. Diagnosed with other mental disorders, including schizophrenia, bipolar disorder, alcohol or substance abuse/dependence, eating disorders, etc.;
2. Individuals with intellectual disabilities or who are unable to cooperate for other reasons, or those lacking or having incomplete civil capacity during the onset of illness;
3. Suffering from neurological or organic brain diseases (such as stroke, cerebral hemorrhage, brain tumors, Parkinson's disease, epilepsy, etc.) and a history of severe traumatic brain injury;
4. Suffering from conditions with high exercise risk, such as hypertension or heart disease;
5. Currently undergoing systematic psychological therapy;
6. In the 3-minute step test, males with a recovery heart rate more than131 and females with a recovery heart rate more than 140;
7. Physically restricted individuals unable to participate in physical exercise;
8. Physical Activity Readiness Questionnaire (PAR-Q) score ≥ 2;
9. Pregnant women or individuals with contraindications to MRI examinations;
10. Individuals with severe suicidal tendencies or at risk of harming others.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating Scale (HAMD) | Week 4 and 8 of treatment duration
  The outcome is assessed by HAMD-17 Scale.

SECONDARY OUTCOMES:
Change from baseline in THINC-it score | Week 4 and 8 of treatment duration
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | Week 4 and 8 of treatment duration
Response to treatment | Week 4 and 8 of treatment duration
  The reduction rate of HAMD-17 or MADRS score was ≥50%
Clinical Global Impression-Severity of Illness (CGI-S) | Week 4 and 8 of treatment duration
Change from baseline in Hamilton Anxiety Rating Scale (HAMA) | Week 4 and 8 of treatment duration
Change from baseline in Ruminative Responses Scale (RRS) | Week 4 and 8 of treatment duration
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) | Week 4 and 8 of treatment duration
Change from baseline in Connor-Davidson Resilience Scale (CD-RISC) | Week 4 and 8 of treatment duration
Rating Scale for Side Effects (SERS) -Antidepressant | Week 4 and 8 of treatment duration
  Rating Scale for Side Effects (SERS) -Antidepressant
Mood Disorder Questionnaire (MDQ) | Week 4 and 8 of treatment duration
International Physical Activity Questionnaire (IPAQ) | Week 4 and 8 of treatment duration
Biomarkers level | Week 0 and 8 of treatment duration
  CRP, IL-1β, TNF-α, IL-6, IL-8, IL-10 and other immune factors, irisin, neurotrophic factor BDNF, vascular endothelial growth factor VEGF, and insulin growth factor IGF-1, NLRP3, CXCL8, CXCL3, CCL5, etc
Body weight in kilograms | Week 4 and 8 of treatment duration
Body fat rate | Week 4 and 8 of treatment duration
Brain imaging features | Week 0 and 8 of treatment duration
  Acquisition was performed by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hostipal, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No